CLINICAL TRIAL: NCT01421056
Title: A Randomized, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Tolerability of Multiple Dose Regimens of CHF 5074 (200, 400, 600 mg/Day for up to 12 Weeks) and to Explore the Effects on Potential Markers of Clinical Efficacy in Patients With Mild Cognitive Impairment
Brief Title: Evaluation of Safety & Tolerability of Multiple Dose Regimens of CHF 5074 and Exploration of Effects on Potential Markers of Clinical Efficacy in Patients With Mild Cognitive Impairment - Open Label Extension (CT04 OLEP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Organization: Chiesi USA, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCD-1014-PR-0053 OLEP; 2010-024270-19 (EudraCT Number)
Record Dates: First submitted 2011-08-05; First posted 2011-08-22 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHF 5074 1x (Experimental): oral tablet, multidose
  Interventions: Drug: CHF 5074 1x
- CHF 5074 2x (Experimental): oral tablet, multidose
  Interventions: Drug: CHF 5074 2x
- CHF 5074 3x (Experimental): oral tablet, multidose
  Interventions: Drug: CHF 5074 3x

INTERVENTIONS:
Drug: CHF 5074 1x — oral tablet, 1x, once a day in the morning for 24 weeks
  Arms: CHF 5074 1x
Drug: CHF 5074 2x — oral tablet, 1x, once a day in the morning for 4 weeks, followed by oral tablet, 2x, once a day in the morning for 20 weeks
  Arms: CHF 5074 2x
Drug: CHF 5074 3x — oral tablet, 1x, once a day in the morning for 4 weeks, followed by oral tablet, 2x, once a day in the morning for 4 weeks, followed by oral tablet, 3x, once a day in the morning for 16 weeks
  Arms: CHF 5074 3x

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ascending oral doses of CHF 5074 after prolonged administration to patients with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of amnestic or non-amnestic Mild Cognitive Impairment.
* Mini-Mental State Examination score higher than 24 at screening.
* MRI scan of the brain at screening with fluid-attenuation inversion recovery (FLAIR) and T2*-weighted gradient-recalled-echo (GRE) sequences.

Exclusion Criteria:

* Diagnosis of Alzheimer's disease according to the (DSM-IV-TR) or NINCDS-ADRDA criteria.
* Any medical condition that could explain the patients cognitive deficits.
* CT or MRI brain imaging results obtained within 12 months prior to baseline showing evidence of infection, infarction, or focal lesions of clinical significance
* MRI scan at screening showing more than 4 cerebral microhemorrhages (lesions with diameter ≤ 10 mm).
* Geriatric Depression Scale (30-point scale) score > 9 at screening.
* History of stroke.
* Modified Hachinski ischemic scale score > 4 at screening.
* Women of childbearing potential.
* Vitamin B12 or folate deficiency.
* Diagnosis of schizophrenia or recurrent mood disorder (including unipolar and bipolar disorders) within 3 years of screening.
* Current diagnosis of peptic ulcer or gastrointestinal bleeding within the last year and/or chronic inflammatory bowel disease.
* Concomitant use of donepezil at doses > 5 mg/day or other cholinesterase inhibitors (rivastigmine or galantamine) at any dose.
* Concomitant use of memantine at dose > 20 mg/day.
* Concomitant use of psychoactive drugs (sedatives, hypnotics, etc).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose of CHF 5074 after multiple oral once daily administration to patients with mild cognitive impairment | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel S. Ross, MD, Principal Investigator — Memory Enhancement Center of America, Inc.; Gabriella Bottini, Prof., Principal Investigator — Osp. Niguarda Ca Granda
Locations (6):
- United States (4):
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Memory Center of New Jersey, Inc., Monroe Twp, New Jersey
  - Memory Enhancement Center of NJ, Inc., Toms River, New Jersey
  - Senior Adults Specialty Research, Austin, Texas
- Italy (2):
  - Clinica Santa Maria, Div Neurologia, Castellanza
  - Osp. Niguarda Ca'Granda, Dip. Di Neuroscienze, Milan